CLINICAL TRIAL: NCT04753931
Title: Investigation of the Effects of Sensory Training Application in Addition to Bobath Training in Stroke Rehabilitation on Balance, Walking and Trunk Position Sensation
Brief Title: Effects of Sensory Training Application in Addition to Bobath Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUOK
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-03

CONDITIONS: Stroke; Stroke Rehabilitation
Keywords: Stroke Rehabilitation; Bobath; Trunk İmpairment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory Training in addition to Bobath Training (Experimental): Exercises will be applied to the individuals participating in the study 3 days a week, 8 weeks, and 24 sessions in total. Exercises will be applied after the conventional therapy sessions.
  Interventions: Other: Sensory Training in addition to Bobath Training
- Bobath Training (Experimental): Exercises will be applied to the individuals participating in the study 3 days a week, 8 weeks, and 24 sessions in total. Exercises will be applied after the conventional therapy sessions.
  Interventions: Other: Bobath Training

INTERVENTIONS:
Other: Sensory Training in addition to Bobath Training — Trunk-focused exercises will be applied for different senses (tactile, proprioceptive, etc.) in addition to Bobath exercises. Bobath exercises will be determined individually according to the evaluation results. In general, exercises aiming to muscle tone regulation, increase balance, walking, and functionality will be applied. Trunk-focused Bobath exercises will be selected.
  Arms: Sensory Training in addition to Bobath Training
Other: Bobath Training — Bobath exercises will be determined individually according to the evaluation results. In general, exercises aiming to muscle tone regulation, increase balance, walking, and functionality will be applied. Trunk-focused Bobath exercises will be selected.
  Arms: Bobath Training

SUMMARY:
The primary purpose of this study is to investigate the effects of sensory training, which will be applied to the trunk in addition to Bobath-based and trunk-focused exercises on trunk functions, sense, balance and gait. The secondary aim of the study is to investigate the effects of Bobath-based and trunk-focused exercises on trunk functional capacity, balance and gait performance.

Our study consists of two groups: Bobath-based trunk training group and, sensory training group in addition to Bobath-based trunk training. The information of individuals who agree to participate in the study and meet the criteria for admission to the study will be recorded with a demographic information form. The scales, questionnaires and tests determined to evaluate the individual's trunk position sense and functions, balance and walking performance will be applied before and after the study.

DETAILED DESCRIPTION:
According to the definition of the World Health Organization, stroke is a clinical scene that develops due to vascular causes, causes focal or global brain damage, begins acutely, and progresses with neurological symptoms lasting 24 hours or longer. İt is stated that stroke is the third leading cause of disability worldwide. As a result of stroke, sensory disturbances may occur in individuals as well as motor symptoms.

The primary purpose of this study is to investigate the effects of sensory training, which will be applied to the trunk in addition to Bobath-based and trunk-focused exercises on trunk functions, sense, balance and gait. The secondary aim of the study is to investigate the effects of Bobath-based and trunk-focused exercises on trunk functional capacity, balance and gait performance.

Our study consists of two groups: Bobath-based trunk training group and, sensory training group in addition to Bobath-based trunk training. All participants will be randomly distributed (using software at http://www.randomizer.org). First, 12 patients will be included in our study and the total number of patients will be determined by calculating the effect size with the interm analysis to be performed later. Exercises will be applied to the individuals participating in the study 3 days a week, 8 weeks and 24 sessions in total. Exercises will be applied to the individuals after conventional therapy session. The information of individuals who agree to participate in the study and meet the criteria for admission to the study will be recorded with a demographic information form. The scales, questionnaires and tests determined to evaluate the individual's trunk position sense and functions, balance and walking performance will be applied before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* Sub-acute (more than three months) and chronic stroke patients.
* Patients are older than 18 years.
* Patients who can sit and walk independently (including those using a walking aid).

Exclusion Criteria:

* Patients with a total score of 20 or more on the trunk impairment scale.
* Patients with additional neurological and/or orthopedic problems that may affect motor performance and balance.
* Patients with mental problems (Mini-Mental State Examination test score <23).
* Patients with communication problems.
* Recurrent stroke patients.
* Patients aged 85 years and over.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Trunk Impairment Scale | The evaluation will be applied at the beginning of the treatment program.
  This scale aims to evaluate the trunk in patients who have suffered a stroke.
Trunk Impairment Scale | The evaluation will be applied at the end of the 8 weeks treatment program.
  This scale aims to evaluate the trunk in patients who have suffered a stroke.
The Stroke Rehabilitation Assessment of Movement (STREAM) | The evaluation will be applied at the beginning of the treatment program.
  STREAM is a measurement tool used to quantitatively evaluate the recovery of voluntary movement and mobility post stroke. The STREAM is used to assess patient's coordination, functional mobility and range of motion.
The Stroke Rehabilitation Assessment of Movement (STREAM) | The evaluation will be applied at the end of the 8 weeks treatment program.
  STREAM is a measurement tool used to quantitatively evaluate the recovery of voluntary movement and mobility post stroke. The STREAM is used to assess patient's coordination, functional mobility and range of motion.
The Fugl-Meyer Assessment (FMA) | The evaluation will be applied at the beginning of the treatment program.
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
The Fugl-Meyer Assessment (FMA) | The evaluation will be applied at the end of the 8 weeks treatment program.
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Berg Balance Scale | The evaluation will be applied at the beginning of the treatment program.
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.
Berg Balance Scale | The evaluation will be applied at the end of the 8 weeks treatment program.
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.
The Barthel Scale/Index (BI) | The evaluation will be applied at the beginning of the treatment program.
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL).
The Barthel Scale/Index (BI) | The evaluation will be applied at the end of the 8 weeks treatment program.
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL).
The Stroke Specific Quality of Life scale (SS-QOL) | The evaluation will be applied at the beginning of the treatment program.
  The Stroke Specific Quality of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke.
The Stroke Specific Quality of Life scale (SS-QOL) | The evaluation will be applied at the end of the 8 weeks treatment program.
  The Stroke Specific Quality of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke.
Functional Reach Test (FRT) | The evaluation will be applied at the beginning of the treatment program.
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task.
Functional Reach Test (FRT) | The evaluation will be applied at the end of the 8 weeks treatment program.
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task.
2 Minute Walk Test (2MWT) | The evaluation will be applied at the beginning of the treatment program.
  The Two/2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity, particularly for those who cannot manage the longer Six Minute Walk Test (6MWT) or 12 Minute Walk Test.
2 Minute Walk Test (2MWT) | The evaluation will be applied at the end of the 8 weeks treatment program.
  The Two/2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity, particularly for those who cannot manage the longer Six Minute Walk Test (6MWT) or 12 Minute Walk Test.
Mini-Mental State Examination | The evaluation will be applied at the beginning of the treatment program.
  The Mini-mental state examination is used to measure cognitive impairment.
Trunk position sense measurements | The evaluation will be applied at the beginning of the treatment program.
  Trunk position senses measurements will be made in trunk flexion and trunk rotation positions. The reposition error method measures the sense of position.
Trunk position sense measurements | The evaluation will be applied at the end of the 8 weeks treatment program.
  Trunk position senses measurements will be made in trunk flexion and trunk rotation positions. The reposition error method measures the sense of position.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Karaca, M.Sc., Study Chair — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)